CLINICAL TRIAL: NCT05947747
Title: A Phase IIb, Randomized, Double-blinded, Placebo-controlled Study to Evaluate the Safety and Efficacy of Exosomes Overexpressing CD24 to Prevent Clinical Deterioration in Patients With Mild-Moderate ARDS
Brief Title: Safety and Efficacy of EXO-CD24 in Preventing Clinical Deterioration in Patients With Mild-Moderate ARDS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nano24med (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SN1
Record Dates: First submitted 2023-05-31; First posted 2023-07-17 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: ARDS

STUDY DESIGN:
Intervention Model Description: This is a two arms study; one arm will receive 10^10 dose of exosomes overexpressing CD24, and the second arm will receive Placebo dose
Who Masked: Participant
Masking Description: The administrated dose will be unknown to the patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: investigational drug EXO-CD24 at a dose of 10^10 (Experimental): 60 patients who will receive a 5-day treatment with the investigational drug EXO-CD24 at a dose of 10^10
  Interventions: Drug: EXO-CD24
- Group 2: treatment in a clean sterile saline solution (placebo) (Placebo Comparator): 30 patients who will receive a 5-day treatment in a clean sterile saline solution (placebo)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: EXO-CD24 — Twice a day for 5 days, dose 10^10
  Other Names: Exosomes Overexpressing CD24
  Arms: Group 1: investigational drug EXO-CD24 at a dose of 10^10
Other: Placebo — Twice a day for 5 days
  Arms: Group 2: treatment in a clean sterile saline solution (placebo)

SUMMARY:
This is phase IIb, Randomized, Double-blinded, Placebo-controlled Study to Evaluate the Safety and Efficacy of Exosomes Overexpressing CD24 of one dose 10^10 exosome particles, to Prevent Clinical Deterioration in Patients with Mild-Moderate ARDS

DETAILED DESCRIPTION:
The study population will include patients with mild-moderate ARDS and laboratory markers predictive of the cytokine storm, who have provided an informed consent.

90 patients will be initially screened, randomized and stratified by center in a 2:1 ratio to receive either 1010 exosome particles (60 patients) or placebo (30 patients).

Study drug will be delivered using standard jet nebulizer that produce aerosol particles size of 0.4-4.4 µm.

The exosomes will be diluted in 1.5 ml normal saline for inhalation, administered twice a day (bid) for 5 days

Study treatments will be given as an add-on to the standard of care. Following the 5 days of treatment, patients will remain in follow-up for 23 additional days. In case of hospital discharge before the full follow-up planned, the patient will be required to return to the site for completion of all study assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Direct and indirect lung injury etiology
2. Age ≥18 years
3. Patients with Early Acute Lung Injury (EALI) > 2 ,or patient on HFNC/NIPPV [(1 point for an oxygen requirement > 2 to 6 liters/min or 2 points for > 6 liters/min; 1 point each for a respiratory rate ≥ 30 breaths/min and baseline immune suppression) (immune system compromised by exogenous drug etc.)] (For saturation goal >90%) [1], or ARDS diagnosis (mild/moderate)
4. Willing and able to sign an informed consent, or has a legal guardian who is able to sign

Exclusion Criteria:

1. Any concomitant illness that, based on the judgment of the investigator might affect the interpretation or the results of the study (immunodeficiency, primary immune deficiency due to virus, hematological malignancy etc.)
2. Patients with SaO2/FiO2<150
3. Patients with mechanical ventilation (ECMO).
4. Pregnancy [positive urine pregnancy test (women of childbearing potential only)] or breastfeeding
5. Participation in any other interventional study in the last 30 days or within 5 half-lives of receiving an investigational agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Safety: Number of participants with treatment-related adverse events as assessed by CTCAE v.5 during the 28 days of the study. | 28 days
Efficacy: the rate of hypoxemic respiratory failure (reported as S/F<150) at day 7 | 7 days
Efficacy: the rate of hypoxemic respiratory failure (reported as S/F<150) at day 28 | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No